CLINICAL TRIAL: NCT07037849
Title: Effects of Control Strategies in Wearable Lower Limb Rehabilitation Robots
Brief Title: The Effects of the Control Strategies of Wearable Lower Limb Rehabilitation Robots
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202421602; U21A20136 (Other Grant/Funding Number: The National Natural Science Foundation of China)
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Gait Training; Gait Disorders
Keywords: Robots; Assistive robots; Trajectory; Torque; Force; Robot kinematics; Knee; Limb; Muscles; Hip
MeSH Terms: conditions — Stroke; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robot gait training group (Experimental): During this study, we will explore which control strategy: Aware Hip Knee Coupling Control (AHKC), Passive control (PC), or fixed compliance control (FCC) may be optimal for post-stroke subjects
  Interventions: Device: Robot-assisted overground gait training

INTERVENTIONS:
Device: Robot-assisted overground gait training — Post-stroke patients were required to complete a session of robot-assisted training, which involved nine repetitions of 5-meter overground walking (three trials for each of the three controllers).

SUMMARY:
Post-stroke patients were required to complete a session of robot-assisted training, which involved nine repetitions of 5-meter overground walking (three trials for each of the three controllers) in a rectangular hospital corridor.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients aged between 18 and 75 years. Patients who are medically stable and able to stand and walk independently for at least 10 meters during rehabilitation.

Stroke event occurred at least 3 months ago Patients with impaired lower limb motor function but with some degree of muscle activity in the lower extremities.

Patients without severe cognitive impairment and capable of understanding and following the treatment protocol.

Patients without severe balance or coordination disorders, able to maintain balance and perform gait training with assistive devices.

Patients without lower limb fractures or other serious skeletal issues affecting the lower limbs.

Patients without severe cardiovascular or other serious illnesses and able to tolerate the intensity and duration of rehabilitation therapy.

Patients willing to participate in the study and able to provide written informed consent.

Exclusion Criteria:

Severe cognitive impairment that prevents the patient from understanding or complying with the treatment protocol.

Severe balance or coordination disorders that prevent the patient from maintaining balance and participating in gait training, even with assistive devices.

Other serious motor disorders, such as abnormal muscle tone or ataxia, which may interfere with the effectiveness of rehabilitation therapy.

Active cardiovascular disease or other serious systemic illnesses that may affect the patient's safety or treatment outcomes.

Lower limb fractures or other serious skeletal issues that may impact the suitability and safety of robot-assisted rehabilitation therapy.

Patients currently receiving other rehabilitation or experimental treatments. Patients with skin ulcers, infections, or other severe skin conditions that may interfere with the use and application of robotic devices.

Unexplained discomfort or pain symptoms that may limit the patient's ability to participate in rehabilitation therapy.

Failure to meet other specific inclusion criteria outlined in the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Change in 10 Meter Walk Test from baseline gait speed | Baseline, immediately after intervention
  Gait speed will be assessed by instructing participants to walk at their maximum safe speed. Each participant will start 1 meter before the designated start line and continue walking until 1 meter past the finish line. The time taken to traverse the measured distance will be recorded using a stopwatch to the nearest one hundredth of a second.

SECONDARY OUTCOMES:
Change scores of Lower Extremity Fugl-Meyer Assessment (FMA-LE) | Baseline, immediately after intervention
  The Lower Extremity Fugl-Meyer Assessment (FMA-LE) is a validated, performance-based scale used to evaluate motor function, reflexes, coordination, and movement synergy of the lower limb in stroke patients. The FMA-LE consists of 17 items, each scored on a 3-point ordinal scale (0 = cannot perform, 1 = performs partially, 2 = performs fully), with a total possible score ranging from 0 to 34. Higher scores indicate better lower limb motor function. Assessments will be performed by trained evaluators according to standardized procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Eight affiliated hospital, Sun Yat-Sen University, Shenzhen, Guangzhou, China